CLINICAL TRIAL: NCT01254292
Title: Multicenter, Randomized, Open-label, Parallel-group Study to Evaluate User Satisfaction With and Tolerability of the Low-dose Levonorgestrel (LNG) Intrauterine Delivery System (IUS) With 12 µg LNG/Day Initial in Vitro Release Rate (LCS12) in Comparison to a Combined Oral Contraceptive Containing 30 µg Ethinyl Estradiol and 3 mg Drospirenone (Yasmin®) in Young Women (18-29 Years) Over 18 Months of Use
Brief Title: LCS12 vs Combined Oral Contraceptive (COC) User Satisfaction Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13362; 2010-020181-21 (EudraCT Number)
Record Dates: First submitted 2010-11-22; First posted 2010-12-06 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Contraception
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LCS12 (Skyla, BAY86-5028) (Experimental): Participants received LCS12 (low dose levonorgestrel [LNG] intrauterine delivery system [IUS]) with an initial in vitro release rate of 12 μg LNG per day for 18 months with optional extension to 36 months
  Interventions: Drug: Levonorgestrel IUD (LCS, BAY86-5028)
- EE30/DRSP (Yasmin, BAY86-5131) (Active Comparator): Participants received combined oral contraceptive (COC) tablet Yasmin containing 30 μg ethinyl estradiol (EE) and 3 mg drospirenone (DRSP) for 18 months/19 cycles
  Interventions: Drug: Yasmin (EE30/DRSP, BAY86-5131)

INTERVENTIONS:
Drug: Levonorgestrel IUD (LCS, BAY86-5028) — LCS12 insertion will occur at randomization visit (Visit 2). Duration of study treatment is 18 months with optional extension to 36 months for subjects in this group only.
  Arms: LCS12 (Skyla, BAY86-5028)
Drug: Yasmin (EE30/DRSP, BAY86-5131) — Combined oral contraceptive (COC; Yasmin; 0.03 mg ethinyl estradiol and 3 mg drospirenone); Subjects will start taking COC at / on the day of visit 2 and continue taking one pill / day without any breaks for the entire study duration of 18 months.
  Arms: EE30/DRSP (Yasmin, BAY86-5131)

SUMMARY:
The primary objective of this study is to evaluate user satisfaction and tolerability in young women (18-29 years of age) using the LCS12 compared with young women using a COC (Yasmin) over a period of 18 months. Subjects in the LCS12 arm will be offered continued use of LCS12 for the full, intended duration of use (up to 3 years) by continuing in a optional, extension phase. Safety data only will be collected during the extension phase of the study.

Secondary objectives are to observe the tolerability, discontinuation rates, adverse event profiles, occurrences of unintended pregnancies (including calculation of Pearl Index [PI]), and bleeding profiles with the two birth-control methods. Additionally, data on missed tablets in the combined oral contraceptive (COC) group, and intrauterine delivery system (IUS) expulsions in the LCS12 group will be recorded. In the LCS12 group, physician satisfaction with the IUS inserter, evaluation of the visibility and texture of the removal threads, and evaluation of the visibility of the LCS12 on ultrasound (in a subset of subjects) will be collected. Finally, in the COC group, information will be collected on the psychosocial impact of missed or delayed pill intake.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed and dated the Informed Consent Form (ICF).
* The subject is generally healthy, requesting contraception, and is between 18 and 29 years of age (inclusive) at Screening.
* In the opinion of the investigator, the subject is

  * in good health;
  * without uterine conditions that would preempt insertion of LCS12;
  * without conditions/history that would contraindicate the use of oral contraceptives.
* Subject has normal or clinically insignificant cervical smear (ie, one that does not require further follow up). A cervical smear must be taken at the Screening Visit or a documented normal result has to have been obtained within 6 months of Screening. Subjects with atypical squamous cells of undetermined significance (ASCUS) can be included in the study if they have a Human Papilloma Virus (HPV) deoxyribonucleic acid (DNA) test that, according to the standards of the local laboratory, is negative for high-risk HPV.
* As determined by subject's history, subject has regular (ie, endogenous cyclicity without hormonal contraceptive use) menstrual cycles (length of cycle 21-35 days).
* Subject is willing and able to attend the scheduled study visits and to comply with the study procedures.

Exclusion Criteria:

* Pregnancy or current lactation (less than 6 weeks since vaginal or Cesarean delivery or abortion). Note: Postpartum LCS12 insertions should be postponed until the uterus is fully involuted, and not earlier than 6 weeks after delivery. If involution is substantially delayed, the investigator should consider waiting until 12 weeks postpartum.
* Infected abortion or postpartum endometritis within 3 months prior to the Screening Visit (Visit 1)
* Chronic, daily use of drugs that may increase serum potassium levels, such as nonsteroidal anti-inflammatory drugs (NSAIDs, eg. ibuprofen and naproxen), potassium-sparing diuretics (eg. spironolactone), potassium supplementation, angiotensin converting enzyme (ACE) inhibitors, angiotensin-II receptor antagonists, aldosterone antagonists, and heparin.
* Abnormal uterine bleeding of unknown origin/undiagnosed abnormal genital bleeding
* Any genital infection (until successfully treated)
* Abnormal cervical smear result (see inclusion criteria)
* Acute, current or history of recurrent pelvic inflammatory disease
* Congenital or acquired uterine anomaly or any distortion of the uterine cavity (eg, by fibroids) that, in the opinion of the investigator, would cause problems during insertion, retention, or removal of LCS12.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 567 (Actual)
Dates: Start 2011-01-06 (Actual); Primary Completion 2013-01-08 (Actual); Study Completion 2014-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (89):
- United States (23):
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Tucson, Arizona
  - Grossmont Center for Clinical Research, La Mesa, California
  - La Mesa, California
  - Genesis Center for Clinical Research, San Diego, California
  - San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Visions Clinical Research, Boynton Beach, Florida
  - Boynton Beach, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Boston, Massachusetts
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Lincoln, Nebraska
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Portland, Oregon
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Philadelphia, Pennsylvania
  - Advanced Research Associates, Corpus Christi, Texas
  - Corpus Christi, Texas
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
  - Seattle, Washington
- Austria (19):
  - Ordination Dr. Schmidl-Amann, Sankt Pölten, Lower Austria
  - Sankt Pölten, Lower Austria
  - Dr. Max Stiglbauer, Wiener Neustadt, Lower Austria
  - Wiener Neustadt, Lower Austria
  - Ordination Dr. Trost, Voitsberg, Styria
  - Voitsberg, Styria
  - Landeskrankenhaus Bregenz, Bregenz, Vorarlberg
  - Bregenz, Vorarlberg
  - Praxis Dr. Hannes Kahr, Graz
  - Graz
  - Dr. Bernhard Svejda, Klagenfurt
  - Klagenfurt
  - Ordination Dr. Sator, Tulln
  - Tulln
  - Dr. Brigitte Wiesenthal, Vienna
  - Vienna
  - Dr. Wolfgang Bartl, Vienna
  - Dr. Walter Paulik, Zeltweg
  - Zeltweg
- Belgium (10):
  - Dr. Philip Loquet, Antwerp
  - Antwerp
  - Hôpital Erasme/Erasmus Ziekenhuis, Bruxelles-brussel
  - Bruxelles-brussel
  - Gynaecologen Noord Antwerpen, Ekeren
  - Ekeren
  - UZ Gent, Ghent
  - Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - Leuven
- Germany (27):
  - Praxis Hr. Dr. A. Soder, Ettlingen, Baden-Wurttemberg
  - Ettlingen, Baden-Wurttemberg
  - Praxis Hr. Dr. K. Greven, Hanover, Lower Saxony
  - Hanover, Lower Saxony
  - Evangelisches Krankenhaus Köln Weyertal gGmbH, Cologne, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Praxis Hr. Dr. E. Goeckeler-Leopold, Geseke, North Rhine-Westphalia
  - Geseke, North Rhine-Westphalia
  - Frauenarztpraxis Dr. Robert Hantschel, Dippoldiswalde, Saxony
  - Dippoldiswalde, Saxony
  - Praxis Hr. Dr. U. Kopprasch, Dresden, Saxony
  - Dresden, Saxony
  - Frauenarztpraxis Dr. Bernd Pittner, Leipzig, Saxony
  - Leipzig, Saxony
  - Praxis Fr. C. Burgkhardt, Leipzig, Saxony
  - Praxis f. Gynäkologie und Geburtshilfe, Bernburg, Saxony-Anhalt
  - Bernburg, Saxony-Anhalt
  - Frauenarztpraxis Dr. Wetzel, Blankenburg, Saxony-Anhalt
  - Blankenburg, Saxony-Anhalt
  - Praxis Hr. H. Thelen, Jessen, Saxony-Anhalt
  - Jessen, Saxony-Anhalt
  - Praxis Fr. Dr. A. Braune, Magdeburg, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Praxis Hr. Dr. D. Rautenberg, Hamburg
  - Hamburg
  - Praxis Hr. Dr. K. Peters, Hamburg
  - Praxis Hr. Dr. K. Buehling, Hamburg
- Russia (10):
  - Altai State Medical University, Barnaul
  - Barnaul
  - Scientific Center of family health & human reprod. problems, Irkutsk
  - Irkutsk
  - Instit. of Motherhood & Childhood care n.a. Gorodkov, Ivanovo
  - Ivanovo
  - City Perinatal Center, Novosibirsk
  - Novosibirsk
  - Institute of Obsteric & Gyn., Saint Petersburg
  - Saint Petersburg

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 42 centers across 4 countries in Austria, Belgium, Germany and United States.
Pre-assignment Details: 644 subjects were screened, of which 77 were screen failures and 567 were randomized, 282 subjects to LCS12 and 285 subjects to Yasmin. 279 subjects randomized to LCS12 while 281 subjects randomized to Yasmin received treatment and started comparative phase up to 18 months. 200 subjects randomized to LCS12 entered extension phase up to 36 months.
Period: Comparative Phase
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Started | 282 | 285
Participants Received Treatment | 279 (safety population) | 281 (safety population)
Completed | 227 | 204
Not Completed | 55 | 81
Not completed — Adverse Event | 25 | 25
Not completed — Lost to Follow-up | 3 | 21
Not completed — Pregnancy | 2 | 6
Not completed — Withdrawal by Subject | 20 | 21
Not completed — Protocol Violation | 1 | 2
Not completed — Wish for pregnancy | 4 | 6
Period: LCS12 Extension Phase
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Started | 200 (A total of 200 participants elected to enter this optional Extension Phase.) | 0 (Optional Extension Phase was for LCS12 group only.)
Completed | 163 | 0
Not Completed | 37 | 0
Not completed — Wish for pregnancy | 14 | 0
Not completed — Adverse Event | 9 | 0
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Other unknown | 4 | 0
Not completed — Pregnancy | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131) | Total
Number analyzed (Participants) | 279 | 281 | 560
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.7 (3.0) | 23.9 (3.0) | 23.8 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 279 | 281 | 560
  Male | 0 | 0 | 0
Number of births [Number; unit: Participants]
  0 | 216 | 206 | 422
  1 | 39 | 49 | 88
  2 | 19 | 24 | 43
  3 | 4 | 2 | 6
  4 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Satisfaction Rate at 18 Months (Last Observation Carried Forward, LOCF)
Description: Satisfaction was to be assessed by the subject based on a 5-point Likert item, using the following question: How satisfied are you with the birth control method used during the study? 1. Very satisfied 2. Satisfied 3. Neither satisfied nor dissatisfied 4. Dissatisfied 5. Very dissatisfied The overall satisfaction rate was to be the percentage of subjects selecting "1. Very satisfied" or "2. Satisfied" for the above question.
Time Frame: At 18 months
Population: Full analysis set (only subjects with at least one assessment of the overall satisfaction rating)
Measure: Number; unit: Percentage of participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 274 | 260
Percentage of participants | 82.1 | 81.9
Statistical Analysis 1: Comparison: LCS12 (Skyla, BAY86-5028); Test type: Superiority or Other; single proportion = 82.1, 95% CI 2-sided [77.1 to 86.5] — Clopper Pearson Confidence Interval
Statistical Analysis 2: Comparison: EE30/DRSP (Yasmin, BAY86-5131); Test type: Superiority or Other; single proportion = 81.9, 95% CI 2-sided [76.7 to 86.4] — Clopper Pearson Confidence Interval

2. Secondary Outcome: Overall Satisfaction Rating by the 5-point Likert Item at 6 Months
Description: as for outcome 1
Time Frame: At 6 months
Population: Full analysis set (only subjects with an assessment of overall satisfaction rating at 6 months)
Measure: Number; unit: Percentage of participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 273 | 260
Percentage of participants
  Very Satisfied | 60.4 | 48.1
  Satisfied | 27.5 | 35.8
  Neither satisfied nor dissatisfied | 7.3 | 9.6
  Dissatisfied | 1.8 | 6.2
  Very Dissatisfied | 2.9 | 0.4

3. Secondary Outcome: Overall Satisfaction Rating by the 5-point Likert Item at 12 Months
Description: as for outcome 1
Time Frame: At 12 months
Population: Full analysis set (only subjects with an assessment of overall satisfaction rating at 12 months)
Measure: Number; unit: Percentage of participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 253 | 238
Percentage of participants
  Very Satisfied | 66.8 | 45.0
  Satisfied | 22.9 | 44.1
  Neither satisfied nor dissatisfied | 5.9 | 5.9
  Dissatisfied | 4.3 | 3.8
  Very Dissatisfied | 0.0 | 1.3

4. Secondary Outcome: Overall Satisfaction Rating by the 5-point Likert Item at 18 Months
Description: as for outcome 1
Time Frame: At 18 months
Population: Full analysis set (only subjects with an assessment of overall satisfaction rating at 18 months)
Measure: Number; unit: Percentage of participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 235 | 217
Percentage of participants
  Very Satisfied | 64.3 | 52.5
  Satisfied | 25.1 | 37.8
  Neither satisfied nor dissatisfied | 6.4 | 6.9
  Dissatisfied | 3.0 | 2.8
  Very Dissatisfied | 1.3 | 0.0

5. Secondary Outcome: Overall Satisfaction Rating by the 5-point Likert Item at End of Study (EOS)
Description: Satisfaction was to be assessed by the subject based on a 5-point Likert item, using the following question: How satisfied are you with the birth control method used during the study? 1. Very satisfied 2. Satisfied 3. Neither satisfied nor dissatisfied 4. Dissatisfied 5. Very dissatisfied The overall satisfaction rate was to be the percentage of subjects selecting "1. Very satisfied" or "2. Satisfied" for the above question.
  The 18-month Treatment Visit served as the End-of-Study (EOS) Visit for participant in the COC group and LCS12 participant who did not enter the Extension Phase.
Time Frame: At 18 months/EOS
Population: Full analysis set (only subjects with an assessment of overall satisfaction rating at 18 months/end of study)
Measure: Number; unit: Percentage of participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 268 | 251
Percentage of participants
  Very Satisfied | 58.6 | 46.6
  Satisfied | 23.5 | 35.1
  Neither satisfied nor dissatisfied | 8.6 | 9.6
  Dissatisfied | 5.6 | 7.6
  Very Dissatisfied | 3.7 | 1.2

6. Secondary Outcome: Overall Satisfaction Rate at 6 Months (LOCF)
Description: as for outcome 1
Time Frame: At 6 months
Population: Full analysis set (only subjects with an assessment of overall satisfaction rating at 6 months or before)
Measure: Number; unit: Percentage of participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 273 | 260
Percentage of participants | 87.9 | 83.8

7. Secondary Outcome: Overall Satisfaction Rate at 12 Months (LOCF)
Description: as for outcome 1
Time Frame: At 12 months
Population: Full analysis set (only subjects with an assessment of overall satisfaction rating at 12 months)
Measure: Number; unit: Percentage of participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 274 | 260
Percentage of participants | 84.3 | 83.8

8. Secondary Outcome: User Satisfaction - Acceptability of the Administration of Study Treatment
Description: The 18-month Treatment Visit served as the End-of-Study (EOS) Visit for participant in the COC group and LCS12 participant who did not enter the Extension Phase.
Time Frame: At 18 months/EOS
Population: Full analysis set (only subjects with an assessment of this questions of the user satisfaction questionnaire at 18 months/end of study)
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 263 | 250
Participants
  Acc. without inconvenience/discomfort | 153 | 186
  Acc. with some inconv/discomfort | 87 | 46
  Not acc. with moderate inconv./discomf. | 11 | 15
  Not acc. with extreme inconv./discomf | 12 | 3

9. Secondary Outcome: User Satisfaction - Choices Upon Completion of the Study
Description: as for outcome 8
Time Frame: At 18 months/EOS
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 263 | 248
Participants
  Continue with study treatment | 174 | 122
  Use a different hormonal contraceptive | 34 | 51
  Use a different contraceptive method | 17 | 27
  Discont. use of all types of contracept. | 6 | 14
  No need for contraceptive at this time | 5 | 12
  Undecided | 27 | 22

10. Secondary Outcome: User Satisfaction - Amount of Menstrual Bleeding
Description: as for outcome 8
Time Frame: At 18 months/EOS
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 260 | 250
Participants
  Decreased | 80 | 35
  Not Changed | 163 | 207
  Increased | 17 | 8

11. Secondary Outcome: User Satisfaction - Satisfaction With Menstrual Bleeding Pattern
Description: as for outcome 8
Time Frame: At 18 months/EOS
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 263 | 250
Participants
  Very satisfied | 101 | 91
  Somewhat satisfied | 65 | 84
  Neither satisfied nor dissatisfied | 48 | 68
  Dissatisfied | 19 | 4
  Very dissatisfied | 10 | 1
  Not applicable | 20 | 2

12. Secondary Outcome: User Satisfaction - Frequency of Experiencing Unexpected Bleeding
Description: as for outcome 8
Time Frame: At 18 months/EOS
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 263 | 250
Participants
  Never | 145 | 219
  Seldom | 92 | 25
  Often | 17 | 5
  Very Often | 9 | 1

13. Secondary Outcome: User Satisfaction - Satisfaction With Menstrual Bleeding Absence
Description: as for outcome 8
Time Frame: At 18 months/EOS
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 130 | 14
Participants
  Very satisfied | 96 | 6
  Somewhat satisfied | 18 | 0
  Neither satisfied nor dissatisfied | 14 | 8
  Dissatisfied | 1 | 0
  Very dissatisfied | 1 | 0

14. Secondary Outcome: User Satisfaction - Comparison of Menstrual Pain Intensity Between Now and Before Treatment
Description: as for outcome 8
Time Frame: At 18 months/EOS
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 259 | 247
Participants
  Decreased | 118 | 61
  Not changed | 102 | 169
  Increased | 39 | 17

15. Secondary Outcome: User Satisfaction - Rating of Usual Menstrual Pain Intensity
Description: as for outcome 8
Time Frame: At 18 months/EOS
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 261 | 249
Participants
  None | 124 | 82
  Mild | 78 | 92
  Moderate | 43 | 67
  Severe | 16 | 8

16. Secondary Outcome: EVAPIL-R Scores at Screening - Composite Score
Description: The EVAPIL-R scale is a self-questionnaire aimed to assess tolerability of oral contraceptives. A composite score was derived from 16 items and the ratings for presence/absence (rated as 1/0), frequency (rated with values from 0 to 2), intensity (rated from 1 to 3) and bother (rated from 1 to 4) for each item. To calculate the composite score, the bother rating of each item was multiplied by an item- specific multiplier and a weight. Range is 0-12, with higher values indicating more severe symptoms/less tolerability.
Time Frame: At screening
Population: Full analysis set (only subjects with an assessment of the EVAPIL questionnaire at screening where the composite score could be calculated)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 273 | 275
Scores on a scale | 0.9386 (0.8036) | 0.8846 (0.8231)

17. Secondary Outcome: EVAPIL-R Scores at Screening - Bother Score
Description: The EVAPIL-R scale is a self-questionnaire aimed to assess tolerability of oral contraceptives. A composite score was derived from 16 items and the ratings for presence/absence (rated as 1/0), frequency (rated with values from 0 to 2), intensity (rated from 1 to 3) and bother (rated from 1 to 4) for each item. To calculate the composite score, the bother rating of each item was multiplied by an item- specific multiplier and a weight. Range is 0-12, , with higher values indicating more severe symptoms/less tolerability.
Time Frame: At screening
Population: Full analysis set (only subjects with an assessment of the EVAPIL questionnaire at screening where the bother score could be calculated)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 273 | 276
Scores on a scale | 0.5569 (0.4451) | 0.5188 (0.4406)

18. Secondary Outcome: EVAPIL-R Scores at 6 Months
Description: as for outcome 16
Time Frame: At 6 months
Population: Full analysis set (only subjects with an assessment of the EVAPIL questionnaire at 6 months where the scores could be calculated)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 252 | 243
Scores on a scale
  Composite score | 1.3187 (0.9888) | 1.1537 (0.9947)
  Bother score | 0.7364 (0.4940) | 0.6550 (0.5148)

19. Secondary Outcome: EVAPIL-R Scores at 12 Months - Bother Score
Description: as for outcome 16
Time Frame: At 12 months
Population: Full analysis set (only subjects with an assessment of the EVAPIL questionnaire at 12 months where the bother score could be calculated)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 233 | 218
Scores on a scale | 0.7789 (0.5120) | 0.6015 (0.4663)

20. Secondary Outcome: EVAPIL-R Scores at 12 Months - Composite Score
Description: as for outcome 16
Time Frame: At 12 months
Population: Full analysis set (only subjects with an assessment of the EVAPIL questionnaire at 12 months where the composite score could be calculated)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 229 | 218
Scores on a scale | 1.4022 (1.0126) | 1.0535 (0.8698)

21. Secondary Outcome: EVAPIL-R Scores at 18 Months/EOS
Description: The EVAPIL-R scale is a self-questionnaire aimed to assess tolerability of oral contraceptives. A composite score was derived from 16 items and the ratings for presence/absence (rated as 1/0), frequency (rated with values from 0 to 2), intensity (rated from 1 to 3) and bother (rated from 1 to 4) for each item. To calculate the composite score, the bother rating of each item was multiplied by an item- specific multiplier and a weight. Range is 0-12, with higher values indicating more severe symptoms/less tolerability. The 18-month Treatment Visit served as the End-of-Study (EOS) Visit for participant in the COC group and LCS12 participant who did not enter the Extension Phase.
Time Frame: At 18 months/EOS
Population: Full analysis set (only subjects with an assessment of the EVAPIL questionnaire at 18 months/end of study where the scores could be calculated)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 260 | 250
Scores on a scale
  Composite score | 1.4804 (1.1926) | 1.0246 (0.9546)
  Bother score | 0.8113 (0.5765) | 0.5908 (0.4836)

22. Secondary Outcome: Cumulative Drop-out Rate
Description: The drop-out rate is the amount of participants that could not complete the study for various reasons. Discontinuation rates due to the following reasons and overall discontinuations were calculated: • LCS12 expulsions • Bleeding pattern alterations • Bleeding pattern alterations with increased bleeding (amount) • Bleeding pattern alterations with decreased bleeding (amount) • Adverse Events The analyses described above were also done by parity. Furthermore, overall discontinuation rates were analyzed by Kaplan-Meier analyses and presented as cumulative half-yearly drop-out rates.
Time Frame: Up to 6, 12, 18, 24 and 36 months
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 279 | 281
Percentage of participants
  Up to 6 months | 7.53 | 11.39
  Up to 12 months | 13.26 | 21.71
  Up to 18 months | 18.64 | 27.40
  Up to 24 months | 30.85 | NA — Extension phase was only for LCS12 group
  Up to 36 months | 33.34 | NA — Extension phase was only for LCS12 group

23. Secondary Outcome: Pearl Index (PI)
Description: The Pearl Index was defined as the number of pregnancies per 100 woman years (WYs). Given the assumption that the number of pregnancies follows a Poisson distribution, the Pearl Index thus is the mean of this distribution.
Time Frame: Up to 18, 24, 36 months
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: Pregnancies per 100 women years
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 279 | 281
Pregnancies per 100 women years
  Pearl index up to 18 months | 0.57 [0.07 to 2.05] | 1.82 [0.67 to 3.97]
  Pearl index up to 24 months | 0.67 [0.14 to 1.95] | NA [NA to NA] — Extension phase was only for LCS12 group.
  Pearl index up to 36 months | 0.65 [0.18 to 1.67] | NA [NA to NA] — Extension phase was only for LCS12 group.

24. Secondary Outcome: Compliance Rate for Yasmin Pill Intake
Time Frame: Up to 18 months
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 281
Percentage of participants
  Missing | 2.8
  Compliance <=75% | 2.1
  Compliance >75% | 95.0

25. Other Pre Specified Outcome: Cumulative Number of Participants With Partial or Total Expulsion
Description: Total expulsion is confirmed if the IUS is observed in the vagina, the IUS is not shown in the uterine cavity by ultrasound, and / or the subject confirms that the system was expelled. Partial expulsion is diagnosed if the IUS can be partially seen in the vagina or is displaced in the cervical canal.
Time Frame: Up to 18, 24, 36 months
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028)
Number analyzed (Participants) | 279
Participants
  Partial expulsion up to 18 months | 0
  Total expulsion up to 18 months | 0
  Partial expulsion up to 24 months | 1
  Total expulsion up to 24 months | 0
  Partial expulsion up to 36 months | 1
  Total expulsion up to 36 months | 0

26. Other Pre Specified Outcome: Investigator's Evaluation of Successful IUS Insertion Procedure
Time Frame: Up to 18 months
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028)
Number analyzed (Participants) | 279
Participants
  Easy | 247
  Slightly difficult | 31
  Very difficult | 1

27. Other Pre Specified Outcome: Participants' Evaluation of Pain During Successful IUS Insertion Procedure
Time Frame: Up to 18 months
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028)
Number analyzed (Participants) | 279
Participants
  None | 49
  Mild | 125
  Moderate | 80
  Severe | 25

28. Other Pre Specified Outcome: Investigator's Evaluation of IUS Removal Procedure
Time Frame: Up to 36 months
Population: Full analysis set (only subjects in the LCS12 arm with documented removal of the IUS)
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028)
Number analyzed (Participants) | 267
Participants
  Easy | 252
  Slightly difficult | 11
  Very difficult | 4

29. Other Pre Specified Outcome: Participants' Evaluation of Pain During IUS Removal Procedure
Time Frame: Up to 36 months
Population: Full analysis set (only subjects in the LCS12 arm with documented removal of the IUS)
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028)
Number analyzed (Participants) | 267
Participants
  None | 136
  Mild | 96
  Moderate | 30
  Severe | 5

30. Secondary Outcome: User Satisfaction - Acceptability of the Administration of Study Treatment
Description: The degree of user satisfaction was assessed at the end-of-study visit using an eight item questionnaire. One of the items assessed was acceptability of study treatment which was categorized into the following: acceptable without I/D, acceptable with some I/D, not acceptable with moderate I/D, and not acceptable with extreme I/D.
Time Frame: At 6 months
Population: Full analysis set (only subjects with an assessment of these questions of the user satisfaction questionnaire at 6 months)
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 256 | 244
Participants
  Acc. without inconvenience/discomfort | 163 | 192
  Acc. with some inconv/discomfort | 87 | 48
  Not acc. with moderate inconv./discomf. | 4 | 4
  Not acc. with extreme inconv./discomf. | 2 | 0

31. Secondary Outcome: User Satisfaction - Acceptability of the Administration of Study Treatment
Description: as for outcome 30
Time Frame: At 12 months
Population: Full analysis set (only subjects with an assessment of these questions of the user satisfaction questionnaire at 12 months)
Measure: Number; unit: Participants
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Number analyzed (Participants) | 237 | 220
Participants
  Acc. without inconvenience/discomfort | 152 | 185
  Acc. with some inconv/discomfort | 74 | 33
  Not acc. with moderate inconv./discomf. | 9 | 2
  Not acc. with extreme inconv./discomf. | 1 | 0

ADVERSE EVENTS:
Time Frame: From start of treatment until 36 months/EOS visit.
Arm/Group | LCS12 (Skyla, BAY86-5028) | EE30/DRSP (Yasmin, BAY86-5131)
Serious Adverse Events (participants affected / at risk) | 22/279 | 5/281
Other Adverse Events (participants affected / at risk) | 215/279 | 148/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCS12 (Skyla, BAY86-5028) (N=279) | EE30/DRSP (Yasmin, BAY86-5131) (N=281)
Basedow's disease (Endocrine disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 2
Infectious mononucleosis (Infections and infestations) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nose deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Basedow's disease (Endocrine disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 2
Breast abscess (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nose deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 0
Breast fibrosis (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Breast prosthesis implantation (Surgical and medical procedures) | 1 | 0
Myomectomy (Surgical and medical procedures) | 1 | 0
Mammoplasty (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCS12 (Skyla, BAY86-5028) (N=279) | EE30/DRSP (Yasmin, BAY86-5131) (N=281)
Vertigo (Ear and labyrinth disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 23 | 4
Abdominal pain lower (Gastrointestinal disorders) | 9 | 5
Abdominal pain upper (Gastrointestinal disorders) | 3 | 6
Constipation (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 9
Gastritis (Gastrointestinal disorders) | 4 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 9 | 14
Toothache (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 3 | 8
Irritability (General disorders) | 3 | 1
Pyrexia (General disorders) | 3 | 2
Acute tonsillitis (Infections and infestations) | 4 | 6
Bronchitis (Infections and infestations) | 4 | 4
Cystitis (Infections and infestations) | 17 | 15
Gastroenteritis (Infections and infestations) | 2 | 4
Influenza (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 17 | 14
Sinusitis (Infections and infestations) | 2 | 6
Tonsillitis (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 11 | 5
Vaginal infection (Infections and infestations) | 8 | 7
Vulvitis (Infections and infestations) | 3 | 0
Vulvovaginal candidiasis (Infections and infestations) | 13 | 7
Vulvovaginitis (Infections and infestations) | 2 | 3
Tooth infection (Infections and infestations) | 0 | 3
Vaginitis bacterial (Infections and infestations) | 9 | 3
Vulvovaginal mycotic infection (Infections and infestations) | 8 | 7
Vulvovaginitis streptococcal (Infections and infestations) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Procedural pain (Injury, poisoning and procedural complications) | 10 | 1
Smear cervix abnormal (Investigations) | 5 | 0
Weight decreased (Investigations) | 1 | 3
Weight increased (Investigations) | 7 | 8
Human papilloma virus test positive (Investigations) | 4 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Headache (Nervous system disorders) | 21 | 33
Migraine (Nervous system disorders) | 2 | 5
Depression (Psychiatric disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 0 | 4
Libido decreased (Psychiatric disorders) | 1 | 3
Mood altered (Psychiatric disorders) | 1 | 3
Breast pain (Reproductive system and breast disorders) | 3 | 1
Breast tenderness (Reproductive system and breast disorders) | 3 | 2
Cervical dysplasia (Reproductive system and breast disorders) | 25 | 16
Dysmenorrhoea (Reproductive system and breast disorders) | 48 | 26
Menorrhagia (Reproductive system and breast disorders) | 5 | 5
Metrorrhagia (Reproductive system and breast disorders) | 9 | 1
Ovarian cyst (Reproductive system and breast disorders) | 19 | 0
Pelvic pain (Reproductive system and breast disorders) | 13 | 0
Vaginal discharge (Reproductive system and breast disorders) | 6 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 6 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 6 | 0
Coital bleeding (Reproductive system and breast disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Acne (Skin and subcutaneous tissue disorders) | 30 | 6
Skin disorder (Skin and subcutaneous tissue disorders) | 3 | 0
Wisdom teeth removal (Surgical and medical procedures) | 4 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 21 | 4
Abdominal pain lower (Gastrointestinal disorders) | 12 | 5
Abdominal pain upper (Gastrointestinal disorders) | 3 | 6
Constipation (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 9
Gastritis (Gastrointestinal disorders) | 5 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 9 | 14
Toothache (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 4 | 8
Pyrexia (General disorders) | 3 | 2
Acute tonsillitis (Infections and infestations) | 5 | 6
Bacterial vaginosis (Infections and infestations) | 18 | 3
Bronchitis (Infections and infestations) | 5 | 4
Cystitis (Infections and infestations) | 23 | 15
Ear infection (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 5 | 4
Gonorrhoea (Infections and infestations) | 3 | 0
Influenza (Infections and infestations) | 5 | 3
Nasopharyngitis (Infections and infestations) | 22 | 13
Sinusitis (Infections and infestations) | 3 | 6
Tonsillitis (Infections and infestations) | 7 | 4
Urinary tract infection (Infections and infestations) | 14 | 4
Vaginal infection (Infections and infestations) | 11 | 7
Vaginitis gardnerella (Infections and infestations) | 4 | 1
Vulvitis (Infections and infestations) | 3 | 0
Vulvovaginal candidiasis (Infections and infestations) | 15 | 6
Vulvovaginitis (Infections and infestations) | 4 | 3
Tooth infection (Infections and infestations) | 0 | 3
Chlamydial infection (Infections and infestations) | 3 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 10 | 7
Vulvovaginitis streptococcal (Infections and infestations) | 3 | 0
Vaginitis chlamydial (Infections and infestations) | 3 | 0
Candida infection (Infections and infestations) | 4 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Procedural pain (Injury, poisoning and procedural complications) | 10 | 1
Smear cervix abnormal (Investigations) | 5 | 0
Weight decreased (Investigations) | 3 | 3
Weight increased (Investigations) | 10 | 8
Human papilloma virus test positive (Investigations) | 5 | 3
Chlamydia test positive (Investigations) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 4
Headache (Nervous system disorders) | 26 | 32
Migraine (Nervous system disorders) | 2 | 5
Depression (Psychiatric disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 0 | 4
Irritability (Psychiatric disorders) | 3 | 1
Libido decreased (Psychiatric disorders) | 3 | 3
Mood altered (Psychiatric disorders) | 1 | 3
Breast pain (Reproductive system and breast disorders) | 3 | 1
Breast tenderness (Reproductive system and breast disorders) | 3 | 2
Cervical dysplasia (Reproductive system and breast disorders) | 35 | 16
Dysmenorrhoea (Reproductive system and breast disorders) | 47 | 26
Dyspareunia (Reproductive system and breast disorders) | 4 | 0
Menorrhagia (Reproductive system and breast disorders) | 6 | 5
Metrorrhagia (Reproductive system and breast disorders) | 10 | 1
Ovarian cyst (Reproductive system and breast disorders) | 18 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 4 | 0
Pelvic pain (Reproductive system and breast disorders) | 13 | 0
Vaginal discharge (Reproductive system and breast disorders) | 12 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 8 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 3 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 6 | 0
Coital bleeding (Reproductive system and breast disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Acne (Skin and subcutaneous tissue disorders) | 34 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 3 | 0
Wisdom teeth removal (Surgical and medical procedures) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less